CLINICAL TRIAL: NCT01973374
Title: Sugar Text: A Randomized Controlled Trial of a Text Message Intervention for Women With Diabetes in Pregnancy
Acronym: Sugar Text
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Celeste Durnwald, Assistant Professor, Maternal Fetal Medicine, Department of Obstetrics and Gynecology Director, Penn Perinatal Diabetes Program Director, High Risk Clinic at the Helen O. Dickens Center for Women's Health, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 817181
Record Dates: First submitted 2013-10-24; First posted 2013-10-31 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes in Pregnancy; Gestational Diabetes; Texting Interventions
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Care (No Intervention)
- Text Message Intervention (Experimental): The text message intervention group receives usual prenatal and diabetic care in addition to two text messages per week throughout the pregnancy and a reminder text message prior to the postpartum visit. The text message intervention group also fills out a survey about the intervention after delivery.
  Interventions: Behavioral: Text Message Intervention

INTERVENTIONS:
Behavioral: Text Message Intervention
  Arms: Text Message Intervention

SUMMARY:
Maternal diabetes in pregnancy can negatively impact fetal well-being and contribute to adverse pregnancy outcomes. Much of the morbidity associated with diabetes in pregnancy can be minimized with tight glucose control. A number of studies in non-pregnant populations have highlighted the feasibility, acceptability and efficacy of text messaging interventions for improving diabetic compliance and control. This study will investigate whether a text messaging intervention is feasible and effective in an urban, diabetic, obstetric clinic and whether this intervention can improve compliance with diabetes care, glucose control and pregnancy outcomes. The study will also assess satisfaction with the intervention itself.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-50 years
* Planned delivery at Hospital of the University of Pennsylvania

Exclusion Criteria:

* Gestational age greater than 34 weeks at initial visit in the Penn Perinatal Diabetes Program
* Women who are unable to read English as all text messages will be in English
* Women who do not have a cellular phone capable of receiving text messages as this is the study intervention

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | date of enrollment up to 12 weeks post partum
  Patient satisfaction with the texting intervention as measured by a post-study survey
Compliance with Obstetric and Diabetes Care | OB screening visit through 12 weeks postpartum
  Proportion of prenatal visits attended, proportion of assigned blood glucose logs sent to clinic for review, proportion of assigned blood glucose values checked, compliance with attendance at postpartum visit.

SECONDARY OUTCOMES:
Efficacy measures | Diabetes diagnosis through 12 weeks postpartum
  Measuring the proportion of blood glucose values within the target range each week; mean fasting and postprandial blood glucose values measured weekly; change in hemoglobin A1C (for pregestational diabetics) from initiation of care to the third trimester
Healthcare Utilization Measures | Screening OB visit through 12 weeks postpartum
  Measuring the number of visits to the perinatal evaluation center related to diabetes care and the total number of antepartum hospitalizations.
Maternal Outcomes | Delivery date through 12 weeks postpartum
  Measuring the mode of delivery (spontaneous vaginal, operative vaginal, cesarean section), complications of delivery (shoulder dystocia, postpartum hemorrhage, third and fourth degree lacerations), and length of hospital stay.
Neonatal Outcomes | Neonate delivery through 12 weeks postpartum
  Measuring fetal demise; neonatal death; birthweight; large for gestational age; small for gestational age; APGAR scores; umbilical cord blood gas; NICU admission; respiratory distress; hypoglycemia; hyperbilirubinemia; length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States